CLINICAL TRIAL: NCT05105971
Title: A Phase 1, Multi-Center, Open-Label Dose Escalation Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BAT6026 in Patients With Advanced Solid Tumors
Brief Title: Assessment of Safety and Preliminary Efficacy With BAT6026 in Solid Tumor Patients in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-6026-001-CR
Record Dates: First submitted 2021-10-24; First posted 2021-11-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- BAT6026 0.01mg/kg (Experimental): BAT6026 0.01mg/kg,intervenous infusion,sample size 1
  Interventions: Drug: BAT6026
- BAT6026 0.03mg/kg (Experimental): BAT6026 0.03mg/kg,intervenous infusion,sample size 1
  Interventions: Drug: BAT6026
- BAT6026 0.1mg/kg (Experimental): BAT6026 0.1mg/kg,intervenous infusion,sample size 3~6
  Interventions: Drug: BAT6026
- BAT6026 0.3mg/kg (Experimental): BAT6026 0.3mg/kg,intervenous infusion,sample size 3~6
  Interventions: Drug: BAT6026
- BAT6026 1mg/kg (Experimental): BAT6026 1mg/kg,intervenous infusion,sample size 3~6
  Interventions: Drug: BAT6026
- BAT6026 3mg/kg (Experimental): BAT6026 3mg/kg,intervenous infusion,sample size 3~6
  Interventions: Drug: BAT6026
- BAT6026 6mg/kg (Experimental): BAT6026 6mg/kg,intervenous infusion,sample size 3~6
  Interventions: Drug: BAT6026
- Amplification group (Experimental): BAT6026 10mg/kg,intervenous infusion,sample size 3~6
  Interventions: Drug: BAT6026

INTERVENTIONS:
Drug: BAT6026 — Phase 1 dose titration study from BAT6026 0.01mg/kg to 10mg/kg, then choose a proper dose for amplification study based on DLT result
  Other Names: anti-OX40 monoclonal antibody

SUMMARY:
the main purpose:

* Evaluate the safety and resistance of BAT6026 injection as a single agent in the treatment of patients with locally advanced or metastatic solid tumors Acceptability
* Explore maximum tolerated dose (MTD) or maximum administered dose (MAD) and be phase II or follow-up clinical The study provides recommended doses and reasonable dosing schedules.

Secondary purpose:

* Evaluate the single dose and multiple doses of BAT6026 injection in patients with locally advanced or metastatic solid tumors Pharmacokinetic (PK) characteristics of the drug;
* Evaluate the immunogenicity of BAT6026 injection;
* Evaluate the pharmacodynamic properties of BAT6026 injection;
* Preliminary evaluation of the anti-tumor efficacy of BAT6026 injection.

DETAILED DESCRIPTION:
This study is designed as a phase I clinical trial of multi-center, open, dose escalation, and extended research.

The study mainly evaluates the safety, tolerability and PK characteristics of BAT6026 injection in patients with advanced malignant solid tumors, explores the maximum tolerated dose and preliminary anti-tumor efficacy, and provides a basis for the recommended dose of subsequent clinical trials.

The research is divided into 2 phases:

The first stage: dose escalation study. The safety, tolerability and pharmacokinetic characteristics of BAT6026 were explored using rapid titration and the "3+3" dose escalation rule.

Because the clinical efficacy benefit of a single drug may be limited, from the ethical point of view of exposing fewer subjects to invalid doses, this dose escalation study uses rapid titration and the "3+3" dose escalation rule to explore the safe dose range . A total of 7 (or 8) dose groups are set up, namely the 0.01 mg/kg group, 0.03mg/kg group, 0.1mg/kg group, 0.3mg/kg group, 1mg/kg group, 3mg/kg group, 6mg/kg Group and 10mg/kg group (optional). Among them, the 0.01mg/kg group and the 0.03mg/kg group use accelerated titration Method to increase the dose; 0.1mg/kg group, 0.3mg/kg group, 1mg/kg group, 3mg/kg group, The 6mg/kg group and the 10mg/kg group were studied in dose escalation according to the standard "3+3" rule.

Group/Ascending Method Dose (mg/kg) Group Number of People A/single subject 0.01 1, or 3~6 B/single subject 0.03 1, or 3~6 C/"Standard 3+3" 0.1 3~6 D/"Standard 3+3" 0.3 3~6 E/"Standard 3+3" 1 3~6 F/"Standard 3+3" 3 3~6 G*/"Standard 3+3" 6 3~6 H*/"Standard 3+3" 10 3~6 *Remarks: After the completion of the dose escalation study of groups A to G, after comprehensive assessment of safety and other factors, it may be considered as appropriate whether to add a 10 mg/kg dose group for further tolerability exploration; it can also be discussed with the investigator according to the specific situation. A new dose is selected between the dose that stops climbing and the previous lower dose group, and the experiment is conducted according to the above rules to determine the more accurate maximum tolerated dose.

The dose escalation rules are as follows:

The first two dose groups A and B adopt an accelerated titration dose escalation plan, that is, cohort size=1. First, one case of group A is included. If no ≥ 2 grade toxic reaction related to the study drug is observed, they can directly enter group B for dose escalation. By analogy with this rule ("1+1"), the increase will be accelerated to Group C. If during the accelerated escalation process, once a group has observed a ≥2 level toxic reaction related to the study drug, the accelerated titration dose escalation should be stopped, and two more subjects need to be included in the dose group to be converted to the standard "3+ 3" dose escalation (ie, cohort size=3) mode until MTD or MAD is reached. Starting from Group C, it is adjusted to the standard "3+3" rule of dose increasing mode, the increasing mode is shown in the following table:

Number of people with DLT/number of people in current dose group Decision of dose increase or decrease 0/3 3 new subjects receive the next high-dose group trial 1/3 The current dose group was added to the group with 3 new subjects 1/3 and 0/3 (ie 1/6) 3 new subjects receive the next high-dose group trial

≥2/3 or ≥2/6 indicates that the dose has exceeded the MTD, and the dose escalation should be stopped. If there are 6 people in the previous dose group, use the previous lower dose group as MTD. If there are only 3 people in the previous dose group, 3 people will be added to the previous dose group. After 3 additional people, if there are ≥ 2 DLTs in the previous dose group, the MTD will continue to decrease. If MTD is explored, the sponsor can discuss with the investigator according to the specific situation and select MTD or a dose lower than MTD as the phase II clinical study Recommended dosage. If the MTD is not reached, the sponsor may also discuss with the investigator based on the specific situation, and select a dose of MAD or a dose group below MAD as the recommended dose for the phase II clinical study as appropriate. As the research progresses, the DLT definition can be revised as appropriate based on new clinical findings. Although the adverse events that meet the DLT criteria or other adverse safety information deemed by the researcher to be meaningful outside the DLT evaluation period do not directly affect the dose escalation decision, they need to be taken into account in the final decision on RP2D. The sponsor and investigator will Before the dose is increased, the existing safety, PK (if any), effectiveness and other information should be used to discuss and comprehensively evaluate the decision-making of dose increase or decrease. When tolerability is explored according to the standard "3+3" dose escalation rule, all subjects in the previous dose group must complete a 21-day DLT observation before the next dose group is enrolled in the cohort. In the dose escalation study, a maximum of 2 subjects in each group are allowed to be in the DLT observation period at the same time. Within each dose group, There must be a time interval of at least 24 hours between the administration of the first enrolled subject and the subsequent enrolled subject.

Adjustments for dose reduction are not allowed. The dose is allowed to be increased as appropriate, but extreme caution is required, and at least it needs to be met at the same time: ①The subject has received at least 4 cycles of study drug treatment; ②After discussion between the sponsor and the investigator, it is deemed that the subject has received a higher first-level dose The treatment of the current dose group will bring more clinical benefits; ③The higher-level dose group has passed the follow-up dose escalation study and proved to have not reached the MTD.

The second stage: Dose extension study. Based on the preliminary safety and effectiveness results of the dose escalation study, the investigator and the sponsor decide whether to choose an appropriate dose group for the extended study, further study the safety and clinical effectiveness of BAT6026, and provide a basis for subsequent clinical studies. A study of 2 dose cohorts is planned, and each cohort has no less than 6 subjects for PK study.

The overall research cycle is roughly divided into the screening period, the treatment period, and the follow-up period:

Screening period: -28d~0d, that is, after signing the informed consent form, the screening evaluation can be completed within 28 days; Treatment period: every 3 weeks is a dosing cycle. The study drug is given on the first day of each cycle. Starting from the second cycle, the dosing time window can be ±3 days, but within 72 hours before each dosing, except In addition to imaging examinations, subjects must complete various examinations including vital signs, laboratory examinations, and physical status scoring. The test subjects also need to complete the clinical tumor imaging evaluation (evaluation The method is consistent, CT or MRI). Study drug treatment should continue until emergence: disease progression/death, or withdrawal due to intolerable toxicity, or acceptance of new anti-tumor therapy due to no therapeutic benefit, or withdrawal of informed consent and voluntary withdrawal for other reasons, or up to 17 Cycles (approximately 1 year), whichever comes first.

The DLT evaluation period is defined as the first treatment cycle, that is, from the first administration to 21 days after the administration.

Follow-up period: If the subject stops using study medication, the treatment period will be deemed to be over(End of Therapy, EOT). All subjects, including those who discontinued treatment for any reason (except for loss of follow-up, death,withdrawal of informed consent), will arrange an EOT visit in a timely manner within 21 + 7 days after receiving the last study drug or before receiving subsequent new anti-tumor treatments . The EOT visit should include vital signs, physical examination, laboratory examination, clinical tumor imaging evaluation (CT or MRI) and other examinations.

Safety follow-up: After receiving the last dose of study drug, the subjects are required to be at 21 + 7 days,A safety visit was conducted on days and 90 days (±7 days), including immune-related adverse events (irAE), until 90 days or the subject received new anti-tumor therapy. Safety visits must be conducted at the research center, and various examinations such as vital signs, physical examinations, and laboratory examinations should be performed to evaluate AEs, concomitant medications, and concomitant treatments. Until the adverse event related to the study drug disappears (or drops to ≤1 level), if the adverse event still exists after the subject stops treatment, the investigator has the discretion to determine the frequency of follow-up according to the actual clinical situation until the investigator considers it undesirable The outcome of the event is returning to normal, stable at an acceptable level, or no further improvement. Survival follow-up: After the safety follow-up, the subjects were followed up for survival every 12 weeks (±14 days), followed by telephone until death, loss of follow-up, withdrawal of informed consent, observation for 1 year or termination of the study.

Subjects will be informed that the sponsor will not provide additional study drugs after completion/discontinuation of study drugs. If necessary, the subjects are recommended to return to the research center, and the investigator and the sponsor will discuss and formulate a new study medication treatment plan for the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years of age ≤75 years of age, gender: men and women are not limited;
2. The investigator estimates that the expected survival period is at least 3 months;
3. The Eastern Cooperative Oncology Group (ECOG) performance status scoring requirement is 0 or 1;
4. Patients with locally advanced or metastatic solid tumors diagnosed by pathology who have failed standard treatment or have no effective treatment methods (refer to CSCO guidelines in 2021);
5. According to the tumor efficacy evaluation standard RECIST 1.1, there must be at least one measurable tumor lesion during the dose expansion stage;

Exclusion Criteria:

1. Have received anti-OX40 monoclonal antibody or double-antibody drug therapy with anti-OX40 activity in the past;
2. It is receiving or expected to receive other anti-tumor treatments during the first study drug administration, including but not limited to chemotherapy, radiotherapy, immunotherapy, hormone therapy (except alternative therapies), targeted therapy, biological therapy, and anti-tumor effects Chinese patent medicine, etc.;
3. Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks before using the study drug for the first time, except for the following items:? Nitrosourea or Mitomycin C is within 6 weeks before the first use of the study drug;? Oral fluorouracil and small molecule targeted drugs are 2 weeks before the first use of the study drug or 5 half-lives of the drug (whichever is longer);? Chinese medicine with anti-tumor indications should be within 2 weeks before the first use of the study drug;
4. Clinical investigators who are participating in this study or who have participated in experimental drugs or medical devices within 4 weeks before the first administration of this study cannot be included;
5. Have been vaccinated within 4 weeks before the first administration or plan to vaccinate live/attenuated vaccines and mRNA vaccines during the study period;
6. Pregnant or lactating women;
7. Patients whose AEs caused by the original anti-tumor therapy within 4 weeks before the first administration of the study drug did not return to CTCAE 5.0≤1 (except for hair loss and fatigue ≤2); previous irAE ≥3 or any level of irAE Those who have terminated immunotherapy;
8. Major surgery (defined as grade 3 and 4 surgery) within 4 weeks before the first administration;
9. Those who have a history of tissue or organ transplantation;
10. Subjects who have had serious infections within 4 weeks before the first administration, including but not limited to infectious complications that require hospitalization, bacteremia, severe pneumonia, etc.; subjects with active infections before the first administration are excluded By;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicity (DLT) | 3 weeks
  safety and tolerability endpoint
maximum tolerated dose (MTD) | 3 weeks
  maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Maximum serum drug concentration（Cmax) | no more than 52 weeks
  pharmacokinetic endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China